CLINICAL TRIAL: NCT05368883
Title: Comparison of the Effects of One-Legged and Two-Legged Exercise Training on Exercise Capacity and Fatigue in Patients With Sarcoidosis
Brief Title: Comparison of Different Exercise Training on Exercise Capacity and Fatigue in Patients With Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tuğçe Tahmaz, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cerrahpasa University
Record Dates: First submitted 2022-04-22; First posted 2022-05-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Sarcoidosis
Keywords: fatigue; exercise; quality of life; pulmonary sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-legged cycling ergometer training (Experimental): One-legged cycling ergometer training; 10 minutes for each leg in the first 2 weeks, 15 minutes of cycling training in the following weeks.
  Interventions: Other: Exercise- One-Legged
- Two-legged cycling ergometer training (Active Comparator): Two-legged cycling ergometer training; 20 minutes for the first 2 weeks, 30 minutes of cycling training in the following weeks.
  Interventions: Other: Exercise-Two-Legged

INTERVENTIONS:
Other: Exercise- One-Legged — The exercise program consisted of a 5-minute warm-up, followed by 10 minutes of cycling for each leg during the first 2 weeks, increasing to 15 minutes for each leg in the subsequent weeks (with a 5-10 minute rest period between switching legs), and concluded with a 5-minute cool-down period. During the exercise, the inactive leg was kept stationary and in contact with the ground . In the one-legged cycling exercise training, whether patients started with the dominant or non-dominant leg was determined randomly
  Arms: One-legged cycling ergometer training
Other: Exercise-Two-Legged — The exercise program consisted of a 5-minute warm-up, followed by 20 minutes of cycling during the first 2 weeks, increasing to 30 minutes in the subsequent weeks, and concluded with a 5-minute cool-down period.
  Arms: Two-legged cycling ergometer training

SUMMARY:
Pulmonary rehabilitation is a key element in the management of people with chronic respiratory disease. A properly followed supervised physical training program in sarcoidosis is safe and has no absolute contraindications. Fatigue can also be associated with sarcoidosis for different reasons. Individualized rehabilitation training can improve the symptoms of patients with sarcoidosis. There is no study in the literature investigating the effectiveness of one-legged exercises that reduce peripheral muscle use, in patients with sarcoidosis. In our study, these two exercise methods will be compared by applying one-legged exercise training and two-legged exercise training. The effect of one-legged exercise training on exercise capacity and fatigue in sarcoidosis patients will be examined. The primary aim of our study is to compare the effects of one-legged exercise training, which is a current exercise approach, and two-legged exercise training on exercise capacity and fatigue in patients with sarcoidosis. The secondary aim is to examine the effect of this exercise training on peripheral muscle strength and quality of life parameters.

DETAILED DESCRIPTION:
Pulmonary rehabilitation is a key element in the management of individuals with chronic respiratory disease. A properly followed supervised physical training program in sarcoidosis is safe and has no absolute contraindications. Fatigue may be associated with different causes in sarcoidosis. Individualized rehabilitation practices can improve the symptoms of patients with sarcoidosis. There is no study in the literature investigating the effectiveness of one-legged exercises that reduce peripheral muscle use in patients with sarcoidosis. In our study, these two exercise methods will be compared by applying one-legged exercise training and two-legged exercise training. 26 patients will be randomly divided into 2 groups (n1=n2=13). While one group will receive one-legged cycling ergometer training, the other group will receive two-legged cycling ergometer training. After 8 weeks of exercise training, patients will be evaluated with, Pulmonary Function Test, Six-Minute Walk Test, Endurance Shuttle Walk test, Fatigue Assessment Scale, Multidimensional Fatigue Inventory, Blood Lactate Level (with lactate device), Medical Research Council Dyspnea Scale, Handheld dynamometer, St. George's Respiratory Questionnaire. The effect of one-legged exercise training on exercise capacity and fatigue in sarcoidosis patients will be examined. The primary aim of our study is to compare the effects of one-legged exercise training, which is a current exercise approach, and two-legged exercise training on exercise capacity and fatigue in patients with sarcoidosis. The secondary aim is to examine the effect of this exercise training on peripheral muscle strength and quality of life parameters. The completion of the study will contribute to the determination of the content of the exercise programs to be applied in sarcoidosis patients and will reveal the effectiveness of one-legged exercise training, which is a current exercise method, in sarcoidosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Disease severity classified as stage 2, 3, or 4 based on chest X-ray findings FAS score ≥ 22 Patients being clinically stable No changes in their medical treatment

Exclusion Criteria:

* Having orthopedic, neurological, cardiac, or metabolic conditions that could hinder participation in the exercise program and adherence to it during the study period.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change of Six-Minute Walking Test Distance from baseline to 8 weeks | 8 weeks
  The distance covered in meters in a straight corridor of 30 meters will be recorded as fast as possible but without running for 6 minutes. The distance that normal individuals should take in this period is 400-700 meters. In addition, oxygen saturation and heart rate, resting fatigue and dyspnea levels will be evaluated with pulse oximetry before and after testing. Modified Borg Dyspnea and Fatigue Scales will be used to determine resting dyspnea and fatigue levels.
Change of Endurance Shuttle Walking Test Distance from baseline to 8 weeks | 8 weeks
  Endurance Shuttle Walk test: This is a standardized field test for the assessment of endurance capacity. In the Endurance Shuttle Walk Test, the participant walks at a constant speed between cones spaced 10 m apart. The selected speed is 85% of the participant's maximum capacity measured in the shuttle walk test at increasing speed. Therefore, before this test, the patient should be given an increasing speed ıncremental shuttle walk test.
Incremental Shuttle Walk Test | 8 weeks
  The incremental shuttle walk test (ISWT) is a field-based assessment of cardiorespiratory fitness and physical function. The ISWT is a performance-based assessment of exercise and functional capacity that measures walking distance in meters. It is a relatively brief and easy test to perform. The ISWT simulates a maximal cardiopulmonary test in a field setting and requires minimal equipment. Longer walking distances signify better performance.

SECONDARY OUTCOMES:
Change of Fatigue Assessment Scale results from baseline to 8 weeks | 8 weeks
  Fatigue Assessment Scale: It includes five-point Likert type options (1=Always-5=Never). Higher scores indicate greater levels of fatigue.
Change of Multidimensional Fatigue Inventory results from baseline to 8 weeks | 8 weeks
  The assessment includes 20 questions that encompass different dimensions of fatigue. These questions are divided into five subscales: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Each subscale consists of 4 questions/statements and employs a 5-point Likert scale. Scores of 53 and above on the questionnaire indicate the presence of fatigue symptoms.
Change of Blood Lactate Level from baseline to 8 weeks | 8 weeks
  To assess fatigue, blood lactate levels, which serve as an objective outcome measure, were taken before exercise, immediately after exercise, at the 5th minute post-exercise, and at the 20th minute post-exercise. A lactate measurement device was used for the blood lactate level measurements. For lactate analysis, a 0.2 μl capillary blood sample was required. Blood samples were taken from the patients' fingertips, placed on the device's strips, and inserted into the designated area of the device. The result was displayed on the device screen in mmol/L within 10 seconds, and the recorded value was noted.

OTHER OUTCOMES:
Dyspnoea | 8 weeks
  The Medical Research Council Scale (MRC) was used to assess dyspnea. The MRC is a five-item scale based on different physical activities that can cause dyspnea. Patients are asked to indicate the level of activity that leads to their dyspnea. The scale rates breathlessness starting from "1," where "1" indicates no dyspnea.
Muscle strength | 8 weeks
  A hand-held dynamometer was used to assess the strength of the quadriceps femoris, tibialis anterior, and gastrosoleus muscles. It has been reported that the hand-held dynamometer is a reliable method for measuring muscle strength.
Health Related Quality of Life | 8 weeks
  Health-related quality of life was assessed using the St. George's Respiratory Questionnaire (SGRQ). The scale has three subdomains: Symptoms (8 items), Activities (16 items), and Impacts of the disease (26 items). The scale score ranges from 0 to 100, with higher scores indicating lower quality of life.
The Leicester Cough Questionnaire (LCQ) | 8 weeks
  The Leicester Cough Questionnaire (LCQ) is an assessment tool used to measure the impact of cough on quality of life and consists of 19 questions. It includes psychological, social, and physical subdomains. Lower scores indicate individuals who are more affected by cough, reflecting a lower quality of life.
Respiratory Function Test | 1. week
  In the current study, the respiratory function test results of patients with sarcoidosis from the past 6 months were recorded. Respiratory function tests (RFT) or pulmonary function tests reflect the physiological characteristics of the lungs (e.g., airflow mechanics, volumes, and gas transfer). RFT measurements are primarily conducted using spirometry. In this study, the participants' RFT measurements were performed using spirometry. Additionally, a diffusion test was conducted for DLCO measurement, an important parameter in interstitial lung diseases. The FEV1, FVC, FEV1/FVC, and DLCO values of the patients were recorded as a result of both measurements. The respiratory function test was conducted in accordance with the ATS/ERS spirometry guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Gökşen KURAN ASLAN, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided